CLINICAL TRIAL: NCT05821348
Title: Salivary Biomarkers of Gastroesophageal Reflux in Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Giorgio Valentina, principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GLORIA
Record Dates: First submitted 2023-03-03; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Gastroesophageal Reflux in Infants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases (Experimental): acting from 2 months up to the first year of life, with age postmenstrual > 40 weeks, hospitalized, with symptoms of GER or GERD and undergoing 24-hour esophageal MII-pH. Saliva samples will be collected during the execution of the MII-pH of the esophagus 24 hours, at defined time points, at least 2 hours after the last meal, so as to study the circadian variations of their composition.
  Interventions: Diagnostic Test: salivary markers
- controls (No Intervention): healthy infants from whom it will be taken a single saliva sample during a health assessment.

INTERVENTIONS:
Diagnostic Test: salivary markers — a description of the salivary biochemical profile of GER infants vs. GERD, so that we can develop non-invasive diagnostic strategies and detect personalized therapeutic treatments.
  Arms: cases

SUMMARY:
Gastroesophageal reflux (GER), defined as the backflow of gastric material into the esophagus, it is a condition with a high prevalence during the first year of life. The disease from Gastroesophageal reflux (GERD), a rarer condition, is defined as the presence of symptoms and complications caused by gastroesophageal reflux. For the diagnosis of GERD in infants it is necessary to perform instrumental diagnostic tests invasive. Several efforts have already been made to identify diagnostic strategies non-invasive but, at the state of the art, no non-invasive biomarker has yet been found of GERD in infants. Therefore, the aim of this pilot study is to identify possible biomarkers salivary gastroesophageal reflux in a population of infants with GER or GERD. Infants from 2 months to the first year of life, with age, will be prospectively enrolled postmenstrual > 40 weeks, hospitalized, with symptoms of GER or GERD and undergoing 24-hour esophageal MII-pH.

Saliva samples will be collected during the execution of the MII-pH of the esophagus 24 hours, at defined time points, at least 2 hours after the last meal, so as to study the circadian variations of their composition.

A control group made up of healthy infants will also be enrolled and will be sampled a single saliva sample during a health assessment. The salivary pH, the buffer capacity, the electrolytes (Na, K, Cl, HCO3) and the saliva pepsin/pepsinogen concentrations of enrolled infants. The expected results include the description of the salivary biochemical profile of GER infants vs. GERD, so that the investigators can develop non-invasive diagnostic strategies and detect personalized therapeutic treatments.

ELIGIBILITY:
Inclusion Criteria:

* Infants with reflux symptoms undergoing MII-pH
* Consent of parents or legal representative

Exclusion Criteria:

* Infants being treated with PPIs
* Infants with postmenstrual age < 40 weeks
* Infants with gastrointestinal disorders/diseases other than functional gastrointestinal disorders (FGID)
* Infants with otorhinolaryngological conditions potentially capable of altering salivary composition
* Infants with gastrointestinal malformations, such as esophageal atresia
* Infants with genetic, neurological, renal or endocrinological disorders
* Infants for whom the collection of salivary samples is not feasible

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
GERD SYMPTOMS | 2 years
  dentify the prevalence of GERD in a cohort of infants with symptoms of gastroesophageal reflux

SECONDARY OUTCOMES:
BIOCHEMICAL PROFILE | 2 years
  Identify any differences in the biochemical profile (pepsin and pepsinogen concentration, electrolyte concentration, such as sodium and HCO3-) of saliva samples collected from healthy, GER and GERD patients.
  Investigate possible circadian variations in the biochemical profile (see above) of saliva samples collected at different "time points" during MII-pH performed in GER and GERD infants Correlate the onset of symptoms and nutrition to any changes in the biochemical profile (see above) of saliva samples taken from GER and GERD infants.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico universitario agostino gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided